CLINICAL TRIAL: NCT01265342
Title: Efficacy Of Nebulised Beclometasone Versus Placebo In Preventing Viral Wheezing In Pre-School Children
Brief Title: Efficacy of Nebulised Beclometasone in Viral Wheezing Prophylaxis
Acronym: ENBe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government); Associazione Culturale Pediatri (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FARM7RANLZ; 2009-011116-38 (EudraCT Number)
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Bronchial Spasm; Respiratory Sounds; Respiratory Tract Infections
Keywords: Bronchial Spasm; Respiratory Tract Infections; Viral wheezing; Child, Preschool; Beclomethasone; Italy; Physicians, Primary Care; Pediatrics
MeSH Terms: conditions — Bronchial Spasm; Respiratory Sounds; Respiratory Tract Infections | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Beclomethasone (Experimental): Beclometasone suspension 400 mcg will be administered through a nebuliser twice a day, in the morning and in the evening, for 10 days
  Interventions: Drug: Beclomethasone

INTERVENTIONS:
Drug: Beclomethasone — Beclomethasone nebulised suspension 400 micrograms twice a day for 10 days
  Arms: Beclomethasone
Drug: Placebo — Placebo nebulised suspension twice a day for 10 days
  Arms: Placebo

SUMMARY:
Inhaled steroids, in particular beclomethasone, are widely prescribed in Italy as symptomatic treatment of upper respiratory infections without evidence of efficacy.

The purpose of this study is to evaluate the efficacy of beclomethasone (administered by nebuliser twice a day) in preventing viral wheezing in pre-school children who had had episodes in the preceding 12 months.

DETAILED DESCRIPTION:
Viral wheezing (intermittent episodes of wheezing induced by viral infection of the upper respiratory tract) is a common condition in pre-school children. Its incidence is estimated between 6 and 30% and varies depending on criteria, diagnosis, and age definition used. Viral wheezing, however, is different from atopic asthma, since in 60% of cases symptoms disappear before the age of 6 . The efficacy of drug treatments in the prevention and/or treatment of viral wheezing is controversial; short acting beta 2 agonists are often considered first choice therapies even if evidence is scarce The usefulness of inhaled steroids is also debated: no benefits are documented for maintenance with low dose inhaled corticosteroids, while their episodic use at a high dose may have a modest improvement in symptoms. Despite the scant evidence, however, nebulised steroids in particular beclomethasone, are widely prescribed in Italy as prophylaxis or treatment for viral wheezing. Beclometasone is the third most prescribed drug in Italian children, with a prevalence estimated around 15% A randomized placebo-controlled trial was therefore planned to evaluate the effectiveness of nebulised beclometasone in preventing viral wheezing in children with upper respiratory tract infections. Besides investigating the drug efficacy, the study could also monitor the incidence of viral wheezing recurrence in preschool children, the disease's natural history and the different therapeutic approaches used by the physicians.

The study will involve 36 Italian family paediatricians from 9 local health units. Children will be randomized to receive beclomethasone or placebo.

The treatment period will last 10 days, and it will be followed by an observational 6 month follow-up period.

Three visits are scheduled: the first at baseline, the second at the end of the treatment period and the third at the end of follow-up period.

During the 10 day treatment period, symptoms will be recorded by the parents on a diary. A clinical evaluation will be performed by the paediatrician during the entry visit and at the end of the treatment period. Moreover, parents will be requested to contact the paediatrician if wheezing occurs during the treatment period and/or the child does not improve within 72 hours from the start of the therapy.

In case of wheezing and/or lack of improvement, paediatricians should visit the child, evaluate the presence of wheezing and rate it. A wheeze score will be assigned as follows: 0 = no wheezing, 1 = end-expiratory wheeze only, 2 = wheeze during entire expiratory with or without inspiratory phase, audible with stethoscope only, 3 = inspiratory and expiratory wheezing audible without stethoscope.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient children 1-5 years old
* Presence of any viral upper respiratory tract infection symptoms
* At least one episode of viral wheezing (diagnosed by a physician) in the last 12 months.
* No, or minimal, asthma-like symptoms in between separate airway infections

Exclusion Criteria:

* Steroid hypersensitivity
* Inhaled and/or oral corticosteroid use in the preceding month
* Chronic respiratory disease (e.g. cystic fibrosis, broncho-pulmonary dysplasia)
* Presence of wheezing at the entry visit

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 576 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
% of children with wheezing (diagnosed by the paediatrician) during the URTI episode.

SECONDARY OUTCOMES:
% of patients needing medical care during the treatment period;
% of patients receiving rescue medication during the treatment period;
% of patients admitted to an emergency department during the treatment period
Duration of the respiratory tract infection episode
% of patients with an asthma-like symptom score (rated by parents) >= 7
Mean asthma-like symptom score for each child
Time to the first viral wheezing episode after the end of the treatment
Frequency of respiratory tract infection episodes during the 6 month follow-up period
Frequency of viral wheezing episodes during the 6 month follow-up period
% of parents who consider the treatment helpful
% of patients fully adherent to therapy
average cost per patient

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Clavenna, MD, Principal Investigator — Mario Negri Institute for Pharmacological Research, Milan, Italy
Locations (9):
- Italy (9):
  - ASL NA/3 Sud, Castellammare di Stabia
  - AUSL Chieti, Chieti
  - ASL Monza Brianza, Monza
  - ASL Torino 3, Pinerolo
  - ASP di Reggio Calabria, Reggio Calabria
  - Ausl Roma E, Roma
  - AUSL Taranto, Taranto
  - Azienda ULSS 20 Verona, Verona
  - ASL 12, Viareggio

REFERENCES:
- [Result] Clavenna A, Sequi M, Cartabia M, Fortinguerra F, Borghi M, Bonati M; ENBe Study Group. Effectiveness of nebulized beclomethasone in preventing viral wheezing: an RCT. Pediatrics. 2014 Mar;133(3):e505-12. doi: 10.1542/peds.2013-2404. Epub 2014 Feb 17. PMID 24534400